CLINICAL TRIAL: NCT04382937
Title: An Open-label, Randomized, Active Control Study to Demonstrate Non-Inferiority in Efficacy, and to Compare Safety and Tolerability of P1101 + Ribavirin to PEG-Intron + Ribavirin in Interferon Treatment-Naïve Subjects With Chronic HCV Genotype 2 Infection
Brief Title: Ropeginterferon Alfa-2b (P1101) Phase 3 Study in Interferon Treatment-Naive Subjects With HCV Genotype 2 Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A14-301
Record Dates: First submitted 2020-04-28; First posted 2020-05-11 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Chronic Hepatitis C Virus Infection
Keywords: P1101; HCV; PEG-Intron
MeSH Terms: interventions — Ribavirin; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P1101 + Ribavirin (Experimental): P1101 400 µg SC Q2W
  Interventions: Drug: P1101 + Ribavirin
- PEG-Intron + Ribavirin (Active Comparator): PEG-Intron 1.5 µg per kg SC Q1W
  Interventions: Drug: PEG-Intron + Ribavirin

INTERVENTIONS:
Drug: P1101 + Ribavirin — P1101 400 µg SC Q2W + Ribavirin 800-1400 mg PO daily
  Other Names: Ropeginterferon alfa-2b
  Arms: P1101 + Ribavirin
Drug: PEG-Intron + Ribavirin — PEG-Intron 1.5 µg per kg SC Q1W + Ribavirin 800-1400 mg PO daily
  Other Names: Peginterferon alfa-2b
  Arms: PEG-Intron + Ribavirin

SUMMARY:
Primary objective:

To demonstrate non-inferiority in sustained virologic response (SVR, undetectable HCV RNA at Follow up week 12) between PEG-Intron 1.5 µg per kg SC Q1W + Ribavirin 800-1400 mg PO daily and P1101 400 µg SC Q2W + Ribavirin 800-1400 mg PO daily for the treatment of chronic HCV genotype 2 infection

DETAILED DESCRIPTION:
Secondary objective:

To determine and compare the efficacy, safety, tolerability and immunogenicity of PEG-Intron 1.5 µg per kg SC Q1W + Ribavirin 800-1400 mg PO daily and P1101 400 µg SC Q2W + Ribavirin 800-1400 mg PO daily

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years of age (or other age required by local regulations); subjects who are over 70 years of age must be in generally good health.
2. Confirmed diagnosis of chronic hepatitis with HCV genotype 2 infection. Chronicity is defined as having proven clinical evidence of chronic hepatitis, e.g. a duration of disease longer than 24 weeks before dosing, OR positive for anti-HCV antibody and HCV RNA at screening with biopsy-proven chronic hepatitis C, OR fibrosis.
3. Compensated liver disease defined by normal or elevated ALT ≤10 x ULN, total bilirubin level <2 mg/dL (except in Gilbert's syndrome), normal albumin, normal INR (INR ≤1.5)
4. Interferon treatment naïve: never received any interferon.
5. No other known form of chronic liver disease apart from chronic hepatitis C infection. But mild and moderate fatty liver diseases can be included.
6. Hemoglobin ≥12 g/dL in men or ≥11 g/dL in women, WBC count ≥3,000/mm3, ANC ≥1,500/mm3, platelet count ≥90,000/mm3; and estimated glomerular filtration rate >60 mL/min.
7. Female and male subjects, and their partners of reproductive potential using effective means of contraception during the whole trial period.
8. Be able to attend all scheduled visits and to comply with all study procedures;
9. Be able to provide written informed consent.

Exclusion Criteria:

Any of the following is cause for exclusion from the study:

1. Decompensated liver disease, including overt clinical symptom and sign of complications related to portal hypertension.
2. Clinically significant illness or surgery within 4 weeks prior to dosing.
3. Any reason which, in the opinion of the investigator, would prevent the subject from participating in the study.
4. Positive test for hepatitis B surface antigen or human immunodeficiency virus at screening.
5. Clinically significant abnormal vital signs at screening.
6. Evidence of severe retinopathy by fundoscopy except age-related macular degeneration at screening.
7. Significant alcohol or illicit drug abuse within one year prior to the screening visit or refusal to abstain from excessive alcohol consumption as defined above or illicit drugs throughout the study.
8. Pregnant or breast feeding female subjects.
9. Therapy with any systemic anti-viral, anti-neoplastic, and immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) within 4 weeks prior to the first dose of study drug.
10. Use of an investigational drug or participation in an investigational drug trial within 4 weeks from the first dose.
11. Known clinically significant presence of any gastrointestinal pathology, clinically significant unresolved gastrointestinal symptoms, clinically significant liver (other than CHC) or clinically significant kidney disease (including but not limited to those with chronic renal failure on dialysis), or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
12. Hospital Anxiety and Depression Scale (HADS) score >10 on depression scale at screening that indicates clinically significant presence of depression determined by investigators.
13. Clinically significant presence of severe neurological disorders, e.g. uncontrolled seizure disorders.
14. Clinically significant presence of severe cardiovascular conditions and severe pulmonary conditions (including but not limited to pulmonary infiltrates, pneumonia, pneumonitis, chronic obstructive lung disease), uncontrolled immunologic, uncontrolled autoimmune, uncontrolled endocrine, uncontrolled metabolic, haematological, severe coagulation disorders or severe blood dyscrasias or other severe uncontrolled systemic disease.
15. A depot injection or an implant of any drug within 3 months prior to administration of study medication, other than contraception or hyaluronic acid injections in joints for osteoarthritis;
16. Body organ transplant and are taking immunosuppressants;
17. History of malignant disease, including solid tumors and hematologic malignancies (except basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured, and carcinoma in situ of cervix); However, subjects who are cancer survivors not on maintenance therapy and who had no malignant diseases history within the past 5 years could be recruited.
18. History of or ongoing opportunistic infection.
19. Serious local infection or systemic infection within the 3 months prior to screening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Subjects with undetectable serum HCV RNA at follow up week 12 | Follow Week 12
  Percentage of subjects with SVR12 (undetectable serum HCV RNA, i.e. <12 IU/mL, at follow up week 12) in each treatment group

SECONDARY OUTCOMES:
Subjects with undetectable serum HCV RNA | Treatment Week 4, 8, 12, 24 and Follow Week 24
  Percentage of subjects with undetectable serum HCV RNA at treatment week 4, 8, 12, 24 (end of treatment) and follow up week 24 in each treatment group
Number of subjects with adverse events | Through study Follow Week 24
  Number of subjects with adverse events in each treatment group
Number of subjects with clinically significant laboratory abnormalities | Through study Follow Week 24
  Number of subjects with clinically significant laboratory abnormalities in each treatment group
Subjects with anti-drug antibodies | Follow Week 12 and 24
  Percentage of subjects with positive anti-drug antibodies (the anti-peginterferon and the anti-Peg) at follow up week 12 and 24
Subjects with neutralizing antibody | Follow Week 12 and 24
  Percentage of subjects with positive neutralizing antibody at follow up week 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Wen Huang, MD/PhD, Study Director — PharmaEssentia
Locations (39):
- China (12):
  - Beijing Ditan Hospital Capital Medical University, Beijing
  - Gansu Wuwei Tumour Hospital, Gansu
  - The First Hospital of Lanzhou University, Gansu
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin
  - Henan Provincial People's Hospital, Henan
  - Luoyang Central Hospital, Henan
  - The First Hospital of Jilin University, Jilin
  - Peace Hospital Affiliated to Changzhi Medical College, Shanxi
  - The Sixth People's Hospital of Shenyang, Shenyang
  - Tangdu Hospital, Fourth Military Medical University, Xi'an
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Xijing Hospital, Fourth Military Medical University, Xi'an
- South Korea (8):
  - Soonchunhyang University Seoul Hospital, Asan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Inha University Medical Center, Incheon
  - Hanyang University Seoul Hospital, Seoul
  - Seoul Metropolitan Government - Seoul National University Boramae Medical Center, Seoul
  - Yonsei University Gangnam Severance Hospital, Seoul
  - Saint Vincent Catholic Hospital, Suwon
- Taiwan (19):
  - Changhua Christian Hospital, Changhua
  - Chang Gung Memorial Hospital, Chiayi Branch, Chiayi City
  - Chia-Yi Christian Hospital, Chiayi City
  - Dalin Tzu Chi Hospital, Chiayi City
  - St. Martin De Porres Hospital, Chiayi City
  - Hualien Tzu Chi Hospital, Hualien City
  - Chang Gung Memorial Hospital, Kaohsiung Branch, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital, Keelung Branch, Keelung
  - Chang Gung Memorial Hospital, Linkou, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Hospital, Liouying, Tainan
  - Chi Mei Medical Center, Tainan
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taitung MacKay Memorial Hospital, Taitung
  - National Taiwan University Hospital Yun-Lin Branch, Yuanlin